CLINICAL TRIAL: NCT00889928
Title: A Trial to Evaluate Natural Orifice Transvaginal Endoscopic Cholecystectomy With Laparoscopic Assistance
Acronym: NOTES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ethicon Endo-Surgery (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CI-08-0004; NCT00821704 (obsolete NCT alias)
Record Dates: First submitted 2009-04-28; First posted 2009-04-29 (Estimated); Results first posted 2011-11-24 (Estimated); Last update posted 2011-11-24 (Estimated); Status verified 2011-11

CONDITIONS: Gallbladder Disease
Keywords: gallbladder disease; cholecystectomy; gallbladder disease indicated for cholecystectomy
MeSH Terms: conditions — Gallbladder Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cholecystectomy (Experimental): transvaginal cholecystectomy
  Interventions: Device: NOTES GEN 1 Toolbox

INTERVENTIONS:
Device: NOTES GEN 1 Toolbox — * Articulating Hook Knife
  * Articulating Snare
  * Articulating Needle Knife
  * Articulating Graspers
  * Articulating Biopsy Forceps
  * Steerable Flex Trocar with Rotary Access Needle
  * Flexible Bipolar Hemostasis Forceps
  * Flexible Maryland Dissector

SUMMARY:
The study will document being able to successfully remove a subject's gallbladder through the vagina (laparoscopic visualization)using a small collection of study surgical tools.

ELIGIBILITY:
Inclusion Criteria

Women will be enrolled in this study who:

1. Are willing to give consent and comply with evaluation and treatment schedule, able to understand and complete study questionnaires;
2. At least 18 years of age;
3. Have a clinical diagnosis of gallbladder disease indicated for cholecystectomy;
4. ASA Classification I or II (Appendix II);
5. Have a negative serum pregnancy test (for women of childbearing potential); and
6. Absence, on visual inspection, of adhesions judged to be a potentially complicating factor in transvaginal access and operation.

Exclusion Criteria

Subjects will be excluded from the study for any of the following:

1. BMI > 35;
2. Use of immunosuppressive medications (within 6 months of surgery; single burst dosages and inhalable steroids are acceptable);
3. Suspicion of gallbladder cancer, tumor, polyps, or mass;
4. Acute cholecystitis or acute pancreatitis;
5. Presence of common bile duct stones;
6. History of cervical or vaginal cancer (or precancerous findings on most recent Pap Test);
7. Pelvic Inflammatory Disease;
8. Evidence of abdominal abscess or mass;
9. Diffuse peritonitis;
10. Use of anticoagulants or anti-platelet agents (use of daily cardio protective doses of aspirin, up to 81 mg/day, is acceptable and shall not constitute an exclusion criterion) or the presence of coagulopathy;
11. Clinical diagnosis of sepsis;
12. History of ectopic pregnancy, pelvic inflammatory disease, or severe endometriosis;
13. History of peritoneal or vaginal trauma;
14. Co-morbid condition(s) that could limit the subject's ability to participate in the study or to comply with follow-up requirements, or that could impact the scientific integrity of the trial;
15. Planned concurrent surgical procedure;
16. Prior or planned major surgical procedure within 30 days before or after study procedure;
17. History of transvaginal surgery;
18. History of (or symptomatic for) abdominal adhesions;
19. Participation in any other investigational device or drug trial that has not completed the primary endpoint or that clinically interferes with the current study endpoints;
20. Previously enrolled in the current series of 4 trials investigating the EES NOTES GEN1 Toolbox;
21. Any contraindication listed in a study device Instructions for Use (IFU) document (if that device may be used in the study procedure); or
22. Any condition which precludes compliance with the study (Investigator discretion).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-04; Primary Completion 2010-11 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hungness, MD, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern University Feinberg School of Medicine - ATTN: Dr Hungness, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cholecystectomy
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cholecystectomy
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 37.7 (6.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Procedure Completion
Description: Completion of procedure - transvaginal removal of the gallbladder
Time Frame: Day of Surgery
Population: All subjects on whom the procedure was attempted.
Measure: Number; unit: participants
Arm/Group | Transvaginal Cholecystectomy
Number analyzed (Participants) | 7
participants | 7

ADVERSE EVENTS:
Arm/Group | Cholecystectomy
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 7/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cholecystectomy (N=7)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Herpes zoster infection neurological (Infections and infestations) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 6 (8)
Urethral injury (Injury, poisoning and procedural complications) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
No significant limitations. Small sample size limits inference to a larger population, however it did allow to assess whether the procedure was feasible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other